CLINICAL TRIAL: NCT01509794
Title: Psychophysiological Indicators of Performance in Computer-Based Simulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Tristan Gorrindo, Co-Director, Division of Post-Graduate Medical Education, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 2011-P-000906
Record Dates: First submitted 2012-01-09; First posted 2012-01-13 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2013-03

CONDITIONS: Healthy
Keywords: CME; Simulation; Affective engagement; Cognitive performance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low Valence (Active Comparator): Participants in the low valence condition will participate in photo-based simulations. They will see a photo of the patient and hear affectively flattened audio. The script and clinical information remain the same as the high valence condition.
  Interventions: Other: Low Valence
- High Valence (Experimental): Participants in the high valence condition will participate in video-based simulations. They will see a rich multimedia presentation of the clinical encounter, with affectively enhanced audio. The script and clinical information remain the same as the low valence condition.
  Interventions: Other: High Valence

INTERVENTIONS:
Other: Low Valence — Participants in the low valence condition will participate in two photo-based simulations: first, an orientation to become familiar with the interface, and then a clinical simulation. Afterward, they will complete a written debriefing followed by an verbal debriefing with a study investigator. They will complete all activities while having their heart rate and galvanic skin response monitored using non-invasive methods.
  Arms: Low Valence
Other: High Valence — Participants in the low valence condition will participate in two video-based simulations: first, an orientation to become familiar with the interface, and then a clinical simulation. Afterward, they will complete a written debriefing followed by an verbal debriefing with a study investigator. They will complete all activities while having their heart rate and galvanic skin response monitored using non-invasive methods.
  Arms: High Valence

SUMMARY:
As simulation is now used in many post-graduate education and assessment domains, the investigators want to learn about how autonomically engaged healthcare providers are with the investigators computer simulation paradigm. The investigators are interested in the relationship between autonomic arousal (as measured by heart rate variability and galvanic skin response), self-report of engagement, and performance in the simulation and cognitive debriefing.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare provider
* Right-handed

Exclusion Criteria:

* Has a medical condition associated with cardiac arrhythmia
* Taking medications (such as antiarrhythmic or beta-blocker) that has an effect on heart rate or autonomic function

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2011-11; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Engagement with simulation | All data will be collected during the one hour when participants engage in the simulation activities and debriefing.
  Participant engagement with simulation will be measured using physiological measures of heart rate variability and galvanic skin response as well as self-report measures during the verbal debriefing.

SECONDARY OUTCOMES:
Cognitive performance | All data will be collected during the one hour when participants engage in the simulation activities and debriefing.
  Cognitive performance will be assessed based on the choices that participants make during the clinical simulation as well as the details that they retain and express during the written debriefing.

CONTACTS AND LOCATIONS:
Overall Officials: Tristan Gorrindo, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Division of Postgraduate Medical Education, Boston, Massachusetts, United States

REFERENCES:
- [Background] Gorrindo T, Baer L, Sanders KM, Birnbaum RJ, Fromson JA, Sutton-Skinner KM, Romeo SA, Beresin EV. Web-based simulation in psychiatry residency training: a pilot study. Acad Psychiatry. 2011 Jul-Aug;35(4):232-237. doi: 10.1176/appi.ap.35.4.232. PMID 21804041